CLINICAL TRIAL: NCT05279001
Title: A Phase 1 Dose Escalation, Safety and Tolerability Study of Jaktinib in Patients With Primary Myelofibrosis (PMF) or Post-polycythemia Vera/Post-essential Thrombocythemia Myelofibrosis (Post-PV/ET MF) and Who Are Relapsed/ Refractory to a Marketed JAK Inhibitor
Brief Title: A Safety and Tolerability Study of Jaktinib
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAKUS001
Record Dates: First submitted 2022-03-02; First posted 2022-03-15 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Jaktinib (Experimental)
  Interventions: Drug: Jaktinib Hydrochloride Tablet

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablet — Orally administered, twice a day

SUMMARY:
This research study is studying a drug called Jaktinib as a possible treatment for Myelofibrosis.

DETAILED DESCRIPTION:
This study is a Phase 1, single-arm, open-label, dose escalation trial, to evaluate the safety and tolerability of Jaktinib in patients with PMF or Post-PV/ET MF and who are relapsed/refractory to a marketed JAK inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelofibrosis (primary, post-polycythemia vera, or post-essential thrombocythemia).
* Relapsed/refractory to a marketed (FDA approved) JAK inhibitor.
* At least 18 years of age.
* ECOG PS 0, 1, or 2.
* Expected life expectancy is greater than 24 weeks.

Exclusion Criteria:

* Any chemotherapy, immunomodulatory therapy, immunosuppressive therapy, corticosteroids, or growth factor treatment within 14 days prior to initiation of study drug.
* Major surgery or radiation therapy within 28 days prior to initiation of study drug.
* With suspected allergies to jaktinib or its excipient.
* Another clinical trial of a new drug or medical instrument within 3 months before screening.
* Females who are pregnant, currently breastfeeding, planning to become pregnant.
* Unable to adopt effective contraceptive methods during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of jaktinib hydrochloride tablets | At least 24 weeks, up to approximately 1 year for follow-up
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Dose-limiting toxicities (DLTs) of jaktinib hydrochloride tablets | 28 days
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Efficacy of jaktinib hydrochloride tablets | at least 24 weeks, up to approximately 1 year
  reduction of spleen volume of ≥35%
Efficacy of jaktinib hydrochloride tablets | at least 24 weeks, up to approximately 1 year
  reduction of total symptoms score (TSS) of ≥50%
Pharmacokinetic characteristics of jaktinib hydrochloride tablets | 7 days
  Peak Plasma Concentration (Cmax)
Pharmacokinetic characteristics of jaktinib hydrochloride tablets | 7 days
  Time to maximum concentration (Tmax)
Pharmacokinetic characteristics of jaktinib hydrochloride tablets | 7 days
  Half-life (T1/2)
Pharmacokinetic characteristics of jaktinib hydrochloride tablets | 7 days
  Clearance (CL/F)
Pharmacokinetic characteristics of jaktinib hydrochloride tablets | 7 days
  Area under Curve (AUCinf)
Pharmacokinetic characteristics of jaktinib hydrochloride tablets | 7 days
  Volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No